CLINICAL TRIAL: NCT01135563
Title: A Phase I Study of Vinblastine and Sirolimus in Pediatric Patients With Recurrent or Refractory Solid Tumors Including CNS Tumors
Brief Title: Study of Vinblastine and Sirolimus in Children With Recurrent/Refractory Solid Tumours Including CNS Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Solving Kids' Cancer (Other)
Responsible Party: Principal Investigator, Sylvain Baruchel, Associate Staff Oncologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000016324
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Solid Tumors; Central Nervous System Tumors
Keywords: pediatrics; Solid Tumors; CNS Tumors; Vinblastine; Sirolimus; Recurrent; Refractory
MeSH Terms: conditions — Central Nervous System Neoplasms; Recurrence | interventions — Vinblastine; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vinblastine and Sirolimus (Experimental): The standard 3+3 Phase 1 trial design will be used for the conduct of this study. Three to six patients can be concurrently enrolled onto a dose level. Accrual is suspended when a cohort of three has been enrolled until toxicity data for that cohort have been reported, or when the study endpoints have been met.
  Interventions: Drug: Vinblastine and Sirolimus

INTERVENTIONS:
Drug: Vinblastine and Sirolimus — Patients will be enrolled to receive vinblastine and sirolimus in 28 day cycles. Using the 3+3 standard Phase1 design, vinblastine will be administered via IV push on Days 1, 8, 15, 22. The starting dose of 4 mg/m2 (Dose Level 1) is 67% of the established MTD (6 mg/m2) for this schedule in pediatrics. Dose escalation will take place in a standard 3+3 design, in which doses will increase by approximately 20 to 25% in successive 3-patient cohorts.
  Sirolimus (rapamycin) will be given by mouth (tablet or suspension) once daily throughout the cycle. Ideally patients will remain on the same dose form (tablet or suspension) for the duration of the study. All patients will be assigned a target sirolimus serum trough
  Other Names: Vinblastine Sulfate Injection; Rapamune

SUMMARY:
This study is a Phase I study using vinblastine and sirolimus in patients with relapsed solid tumors including selected brain tumors and lymphoma. The investigators hypothesis is that the combination administration of weekly vinblastine and sirolimus is safe.

DETAILED DESCRIPTION:
Published data demonstrating a survival advantage of the vinblastine-sirolimus regimen vs single agent in an orthopotic neuroblastoma mouse model and our unpublished data support a VBL in vitro pro-apoptotic plasma concentration of 1-2 nM range and an anti angiogenic concentration of 2pM. These plasma concentrations are achievable with a 6 mg/m2 (apoptosis) and 1 mg/m2 VBL regimen (anti-angiogenesis) weekly regimen. We expect that vinblastine delivered at any given dose, as described in the protocol, will carry both anti-apoptotic and antiangiogenic activity. Safety and preliminary efficacy of both drugs in pediatric tumors support the development of a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 0-21 years at the time of diagnosis
2. Diagnosis: Histologic verification at either the time of original diagnosis or relapse of solid tumor including CNS tumors or lymphomas
3. Disease Status: All refractory/recurrent solid tumors including CNS tumors (all Diffuse Intrinsic Brain Stem Gliomas excluded) and lymphomas that have relapsed after, or are refractory to, a chemotherapy-containing treatment regimen
4. Measurable disease:

   * Measurable tumor by CT or MRI defined as >10 mm by spiral CT in at least one dimension
5. Current disease state must be one for which there is currently no known curative therapy
6. A negative urine pregnancy test is required for female participants of child bearing potential
7. Organ Function Requirements:

   * adequate liver function as defined by AST or ALT < 5 x upper limit of normal, bilirubin ≤1.5 X upper limit of normal
   * adequate renal function: Serum creatinine < 1.5 X upper limit of normal for age
8. Adequate Bone Marrow Function Defined as:

   * ANC ≥ 1000/mm3, platelets ≥ 75,000/mm3 and hemoglobin ≥ 90 g/L
   * Transfusions are permitted to meet these platelet and Hgb criteria, if the patient is known to have a history of bone marrow involvement with tumor
   * Patients with platelet counts < 75,000/ mm3 who are refractory to platelet transfusions are not eligible for this study
   * Patients requiring transfusions of platelets or RBC to meet eligibility criteria will not be evaluable for platelet or hgb/hct hematological toxicity
9. Lansky Play Score (for patients < 16 years of age) must be more than 50 and/or ECOG performance status (for patients ≥ 16 years of age) must be 0 to 2
10. Specific requirements for Neuroblastoma patients Stratum:

    * MIBG scan with positive uptake at minimum of one site (MIBG not required if subject's neuroblastoma is previously determined to not uptake MIBG and no measurable disease)
    * Bone marrow with tumor cells seen on routine morphology (not by NSE staining only) of bilateral aspirate and /or biopsy on one bone marrow sample
11. Written informed consent

Exclusion Criteria:

1. Lansky score <50%
2. Investigational Drugs: Patients who are currently receiving another investigational drug(s)
3. Previous treatment with Vinblastine and/or mTor inhibitors
4. Anti-cancer Agents: Patients who are currently receiving other anticancer agents. Patients must have fully recovered from the effects of prior chemotherapy, generally at least 3 weeks from the most recent administration (6 weeks for nitrosoureas)
5. Infection: Patients who have an uncontrolled infection are not eligible until the infection is judged to be well controlled
6. Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study, or in whom compliance is likely to be suboptimal
7. One week from usage of hematopoietic Growth Factor
8. Patients who are refractory to platelet transfusions
9. Brain Stem Glioma patients

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2010-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of vinblastine in combination with sirolimus | 12 months
  Maximum tolerated dose (as defined by protocol) of vinblastine in combination with sirolimus

SECONDARY OUTCOMES:
Safety data | 12 months
  Safety data will be described for all patients receiving at least one dose of vinblastine and sirolimus. Safety data will include values for hematology, serum chemistry, vital signs, and adverse events. The proportion of patients experiencing adverse events, serious adverse events, dose limiting toxicities and treatment delays will be summarized for each dosing cohort.
Response Rate | 12 months
  The proportion of patients experiencing progressive disease, stable disease, partial responses or complete responses will be summarized in tabular format. Progression free survival and duration of any responses will also be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Baruchel, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (5):
- United States (3):
  - Rady Children's Hospital-San Diego, San Diego, California
  - SSM Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Fletcher Allen Health Care, Burlington, Vermont
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec

REFERENCES:
- [Background] Morgenstern DA, Marzouki M, Bartels U, Irwin MS, Sholler GL, Gammon J, Yankanah R, Wu B, Samson Y, Baruchel S. Phase I study of vinblastine and sirolimus in pediatric patients with recurrent or refractory solid tumors. Pediatr Blood Cancer. 2014 Jan;61(1):128-33. doi: 10.1002/pbc.24656. Epub 2013 Aug 17. PMID 23956145